CLINICAL TRIAL: NCT03759184
Title: Phase 1 Trial of Human IL-15 (rhIL-15) and Obinutuzumab for Relapsed and Refractory Chronic Lymphocyte Leukemia
Brief Title: Human IL-15 (rhIL-15) and Obinutuzumab for Relapsed and Refractory Chronic Lymphocyte Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was closed after > 1 year of inactivity.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin Conlon, MD, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 190024; 19-C-0024
Record Dates: First submitted 2018-11-28; First posted 2018-11-29 (Actual); Results first posted 2022-03-10 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Leukemia; Lymphocytic; Chronic; B-Cell
Keywords: Monoclonal Antibody Treatment; Recombinant Human Interleukin-15; Lymphoid Malignancy; Antibody-Dependent Cell-Mediated Cytotoxicity (ADCC)
MeSH Terms: conditions — Leukemia; Bronchiolitis Obliterans Syndrome | interventions — Interleukin-15; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 -DOSE ESCALATION (Experimental): DOSE ESCALATION: Interleukin-15 (IL-15) by continuous intravenous (civ) infusion at escalating doses of 0.5, 1, and 2 mcg/kg/day on days 1-5 of each 4-week cycle (max 6 cycles), with Obinutuzumab by IV infusion at a dose of 100 mg on day 4, 900 mg on day 5, 1,000 mg on day 11, and 1,000 mg on day 18 of the first cycle; then 1,000 mg on day 4 of each subsequent cycle, to determine the maximum tolerated dose (MTD)
  Interventions: Drug: rhIL-15; Biological: Obinutuzumab
- Arm 2 - DOSE EXPANSION (Experimental): DOSE EXPANSION: 3 to 6 patients to receive interleukin-15 (IL-15) by continuous intravenous (civ) infusion at the maximum tolerated dose (MTD) on days 1-5 of cycles 1-6 with Obinutuzumab by IV infusion at a dose of 100 mg on day 4, 900 mg on day 5, 1,000 mg on day 11, and 1,000 mg on day 18 of the first cycle; then 1,000 mg on day 4 of each subsequent cycle (Total 9 patients at MTD)
  Interventions: Drug: rhIL-15; Biological: Obinutuzumab

INTERVENTIONS:
Drug: rhIL-15 — Continuous intravenous (civ) Interleukin-15 (IL-15) at dose levels of 0.5,1 or 2 mcg/kg/day on days 1-5 of cycles 1-6
  Other Names: Recombinant human interleukin-15
  Arms: Arm 1 -DOSE ESCALATION
Drug: rhIL-15 — Continuous intravenous (civ) Interleukin-15 (IL-15) at the maximum tolerated dose or the maximum administered dose of 2 mcg/kg/day on days 1-5 of cycles 1-6
  Other Names: Recombinant human interleukin-15
  Arms: Arm 2 - DOSE EXPANSION
Biological: Obinutuzumab — Intravenous (IV) Obinutuzumab will be administered at a dose of 100 mg on day 4, 900 mg on day 5, 1,000 mg on day 11, and 1,000 mg on day 18 of cycle 1: then 1,000 mg on day 4 of each subsequent cycle
  Other Names: Gazyva

SUMMARY:
Background:

Chronic lymphocytic leukemia (CLL) is a blood cancer. Recombinant human interleukin 15 (IL-15) is a manmade protein. Obinutuzumab is a protein made to deactivate cancer cells. Researchers want to see if treating people with CLL with both proteins improves their outcomes.

Objectives:

To find the safe dose of IL-15 with Obinutuzumab. To identify its effects, including on the immune system and cancer.

Eligibility:

Adults at least 18 years old who have certain CLL that standard therapy has failed

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Evaluation of ability to do daily activities
* Blood, heart, and urine tests

Participants may also be screened with:

* A small amount of bone marrow removed by needle in the hipbone
* Scans of the body and/or brain

The study will be done in 28-day cycles for up to 6 cycles.

Participants will get the study drugs through a catheter and pump.

Cycle 1: Participants will be seen in the clinic during week 1. They will get:

* IL-15 as a continuous intravenous infusion over 24 hours on days 1-5 and 3 dose levels will be evaluated: dose level 1; 0.5 mcg/kg/day; dose level 2: 1 mcg/kg/day and dose level 3: 2 mcg/kg/day.
* Obinutuzumab as a 4-hour infusion in escalating doses during the course of the first cycle 100 mg on day 4, 900 mg on day 5, 1000 mg on day 11 and day 18.

Cycles 2 through 6: Participants will come to the clinic days 1-5 and get IL-15 as in cycle 1 and Obinutuzumab 1000 mg on day 4 of each treatment cycle.

During the study, participants:

* Will repeat screening tests
* Will get standard medicines for side effects
* May give blood, saliva, and tumor samples for research

After treatment, participants will have follow-up visits every 3 months for 1 year, then every 6 months for up to 5 years. After that, participants may be called or emailed.

DETAILED DESCRIPTION:
Background:

* Of the several drugs and drug combinations approved for treatment of relapsed and refractory chronic lymphocytic leukemia (CLL), the reported complete response rates are no greater than 30%.
* Obinutuzumab is a glycoengineered, humanized type 2 anti-cluster of differentiation 20 (CD20) monoclonal antibody thought to engage the immune system by directly activating antibody-dependent, cell mediated cytotoxicity (ADCC); it is approved for treatment of chronic lymphocytic leukemia in combination with chlorambucil.
* The key mediators of ADCC are polymorphonuclear neutrophils, monocytes, and natural killer (NK) cells.
* Recombinant human Interleukin-15 (rhIL-15) is a stimulatory cytokine that promotes the differentiation and activation of NK cells, monocytes, and long-term cluster of differentiation 8 (CD8) + memory T-cells. In a Phase I trial, administration of rhIL-15 as a 5-day continuous intravenous infusion (civ) was associated with up to 45-fold increase in the number of NK cells at well tolerated dose levels.
* Preclinical murine lymphoid malignancy models have shown increased efficacy of monoclonal antibodies when administered together with recombinant human Interleukin-15 (rhIL-15); BL/6 mice inoculated with EL4 murine T-cell lymphoma expressing human cluster of differentiation 20 (EL4-CD20) cells (a syngeneic lymphoma line); including significant prolongation of survival with the IL-15/Rituximab combination compared to either drug given as single agent (90% v. 30% alive at 75 days).

Objectives:

- To determine the safety, toxicity profile, dose-limiting toxicity (DLT) and the maximum tolerated dose (MTD) of civ rhIL-15 administration in combination with intravenous (IV) Obinutuzumab treatment

Eligibility:

* Age greater than or equal to 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1
* Diagnosis of chronic lymphocytic leukemia (CLL) with greater than or equal to 50% of B cells expressing CD20
* Patients must have measurable or evaluable disease
* Patients must have CLL that is refractory or relapsed following therapy with a Bruton's tyrosine kinase (BTK) inhibitor OR have relapsed/refractory CLL and are intolerant to BTK inhibitor therapy; patients with deletion 17p (del(17p) must also be refractory or relapsed after, or intolerant to, therapy with Venetoclax
* Adequate organ function parameters as defined within the protocol
* Active disease requiring treatment, as defined within the protocol

Design:

* This is a single institution non-randomized Phase I dose escalation study evaluating increasing doses of civ rhIL-15 in combination with Obinutuzumab using a standard 3 + 3 dose escalation design.
* On days 1-5 of each 4-week cycle, rhIL-15 will be administered by civ at dose levels 0.5, 1, and 2 mcg/kg/day.
* During the first cycle, Obinutuzumab will be administered at a dose of 100 mg by IV on day 4, 900 mg on day 5, 1,000 mg on day 11, and 1,000 mg on day 18: then 1,000 mg on day 4 of each subsequent cycle.
* Infusion reaction, antimicrobial, and tumor lysis syndrome prophylaxis will be administered per manufacturers recommendations.
* Treatment will continue up to 6 cycles, or until unacceptable toxicity or progressive disease.
* Up to 24 patients will be enrolled in the study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have a confirmed diagnosis of chronic lymphocytic leukemia/small lymphocytic lymphoma that expresses cluster of differentiation 20 (CD20) as confirmed by new/fresh peripheral blood sample collection and review by Laboratory of Pathology, National Cancer Institute (NCI)
* Measurable or evaluable disease
* Patients must have received prior treatment required as follows: chronic lymphocyte leukemia (CLL) that is refractory or relapsed following therapy with a Bruton's tyrosine kinase (BTK) inhibitor OR have relapsed/refractory CLL and are intolerant of BTK inhibitor therapy; in addition, patients with deletion 17p (del(17p) must also be refractory or relapsed after, or intolerant to, therapy with Venetoclax; patients who have received prior Obinutuzumab are eligible regardless of response to the drug.
* Active disease requiring treatment, as defined by at least one of the following (per the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2018 consensus criteria):

  * Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia (hemoglobin (Hb) <10 g/dL) and/or thrombocytopenia (platelet counts <100x10^9/L).
  * Massive (i.e., greater than or equal to 6 centimeters (cm) below the left costal margin) or progressive or symptomatic splenomegaly.
  * Massive nodes (i.e., greater than or equal to 10 cm in longest diameter) or progressive or symptomatic lymphadenopathy.
  * Progressive lymphocytosis with an increase of greater than or equal to 50% over a 2-month period, or lymphocyte doubling time (LDT) <6 months.
  * Autoimmune complications including anemia or thrombocytopenia poorly responsive to corticosteroids.
  * Symptomatic or functional extranodal involvement (e.g., skin, kidney, lung, spine).
  * Disease-related symptoms as defined by any of the following:

    * Unintentional weight loss greater than or equal to 10% within the previous 6 months.
    * Significant fatigue (i.e., Eastern Cooperative Oncology Group (ECOG) performance scale 2 or worse; cannot work or unable to perform usual activities).
    * Fevers 38.0 degree Celsius (C) for 2 or more weeks without evidence of infection.
    * Night sweats for greater than or equal to 1 month without evidence of infection.
* greater than or equal to 18 years of age on day of signing informed consent

NOTE: Because no dosing or adverse event data are currently available on the use of rhIL-15 in combination with Obinutuzumab in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials

* ECOG performance status less than or equal to 1 (Karnofsky greater than or equal to 80%; or less than or equal to 2 (Karnofsky >60%) if the decrease in the performance status is CLL-related and constitutes a criterion for active treatment
* Adequate organ function as evidenced by the following laboratory parameters:

  * Absolute neutrophil count (ANC) greater than or equal to 750 /mcL
  * Platelets greater than or equal to 50,000 / mcL (transfusions not permitted)
  * Hemoglobin greater than or equal to 9 g/dL (transfusions permitted)
  * Serum creatinine less than or equal to 1.5 X upper limit of normal (ULN)
  * Serum total bilirubin less than or equal to 1.5 X ULN OR Direct bilirubin less than or equal to upper limit of normal (ULN) for patients with total bilirubin levels > 1.5 ULN
  * Aspartate aminotransferase (AST) Serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) Serum glutamate-pyruvate transaminase (SGPT) less than or equal to 3 X ULN
* Women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study treatment, and for at least 18 months after the last dose of Obinutuzumab. The effects of rhIL-15 and Obinutuzumab on the developing human fetus are unknown. Additionally, CD20-depleting agents are known to produce opportunistic infections, causing fetal B-cell depletion in animal studies, and may be teratogenic. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

NOTE: WOCBP is defined as any female who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal. WOCBP must have a negative pregnancy test (Human chorionic gonadotropin (HCG) blood or urine) during screening.

- Ability of patient to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Current or prior anti-cancer treatment prior to the first dose of rhIL-15 as defined below:

  * Chemotherapy, targeted small molecule therapy, or other anti-cancer treatment not otherwise specified below within 2 weeks
  * Radiation therapy within 2 weeks
  * Anti-cancer monoclonal antibody (mAb) treatment within 4 weeks
  * Use of an investigational agent (e.g., biologic, drug, or other) within 4 weeks
  * Allogeneic stem cell transplant within 100 days
  * Systemic treatment for graft versus host disease (GVHD), including but not limited to oral or parenteral corticosteroids, ibrutinib, and extracorporeal phototherapy, within the last 12 weeks
* Persisting toxicity related to prior therapy (including GVHD) of grade > 1, with the exception of the following: alopecia or sensory neuropathy grade less than or equal to 2, or other grade less than or equal to 2 not constituting a safety risk based on investigator's judgment
* Current use of immunosuppressive medication, EXCEPT for the following:

  * Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection).
  * Systemic corticosteroids at physiologic doses less than or equal to 10 mg/day of prednisone or equivalent; or,
  * Steroids as premedication for hypersensitivity reactions (e.g., computed tomography (CT) scan premedication)
* Presence of Richter's transformation.
* Patients requiring immediate cytoreduction, if they had no prior treatment with a drug that has an established clinical benefit.
* Presence of uncontrolled intercurrent illnesses including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, cognitive impairment, active substance abuse, or psychiatric illness/social situations that in the view of the Investigator would preclude safe treatment and limit compliance with study requirements
* Presence of active bacterial infections, documented human immunodeficiency virus (HIV) infection, polymerase chain reaction (PCR) evidence for active or chronic hepatitis B or hepatitis C, or positive screening hepatitis B virus (HBV)/ hepatitis C virus (HCV) serology without documentation of successful curative treatment
* Asthma requiring chronic inhaled or oral corticosteroids, or history of asthma requiring mechanical ventilation; patients with a history of mild asthma that are on or can be switched to non-corticosteroid bronchodilator regimens are eligible
* Active or history of any autoimmune disease thought to be unrelated to their CLL
* Inability or refusal to practice effective contraception during therapy or the presence of pregnancy or active breastfeeding. Because there is no significant preclinical information regarding the risks to a fetus or a newborn infant, all pregnant or breastfeeding woman will be excluded from participation in this trial
* Received a live vaccine within 30 days of planned start of study therapy. NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to rhIL-15 or Obinutuzumab, unless felt to be in the best interests of the patient in the opinion of the investigator
* Known additional malignancy that requires active systemic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2021-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Conlon, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genome Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research (BTRIS) and with the permission of the study principal investigator (PI).
  Genomic data are made available via database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Derived] Dubois SP, Miljkovic MD, Fleisher TA, Pittaluga S, Hsu-Albert J, Bryant BR, Petrus MN, Perera LP, Muller JR, Shih JH, Waldmann TA, Conlon KC. Short-course IL-15 given as a continuous infusion led to a massive expansion of effective NK cells: implications for combination therapy with antitumor antibodies. J Immunother Cancer. 2021 Apr;9(4):e002193. doi: 10.1136/jitc-2020-002193. PMID 33883258
- [Derived] Waldmann TA, Dubois S, Miljkovic MD, Conlon KC. IL-15 in the Combination Immunotherapy of Cancer. Front Immunol. 2020 May 19;11:868. doi: 10.3389/fimmu.2020.00868. eCollection 2020. PMID 32508818
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0024.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were enrolled on the dose expansion phase of the study because the study was closed after > 1 year of inactivity.
Groups:
- Arm 1 - Dose Escalation - Dose Level 1: Each cycle of treatment is 28 days or 4 weeks, and a maximum of 6 cycles will be administered.
  Participant was treated with continuous intravenous (civ) interleukin-15 (IL-15) on dose level 1 with 0.5 mcg/kg/day on days 1-5 of cycles 1-6.
  Obinutuzumab (IV) will be administered at a dose of 100 mg on day 4, 900 mg on day 5, 1,000 mg on day 11, and 1,000 mg on day 18 of cycle 1: then 1,000 mg on day 4 of each subsequent cycle.
Period: Overall Study
Arm/Group | Arm 1 - Dose Escalation - Dose Level 1
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1 - Dose Escalation - Dose Level 1
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-emergent Adverse Events (AEs) Related to Recombinant Human Interleukin-15 (rhIL-15)
Description: Here is the number of treatment-emergent AEs related to rhIL-15 assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. A treatment emergent AE is defined as
Time Frame: 28 days or 4 weeks (cycle 1)
Measure: Number; unit: adverse events
Arm/Group | Arm 1 - Dose Escalation - Dose Level 1
Number analyzed (Participants) | 1
adverse events | 0

2. Primary Outcome: Number of Treatment-emergent Adverse Events (AEs) Related to Obinutuzumab
Description: Here is the number of treatment-emergent AEs related to Obinutuzumab assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. A treatment emergent AE is defined as
Time Frame: 28 days or 4 weeks (cycle 1)
Measure: Number; unit: adverse events
Arm/Group | Arm 1 - Dose Escalation - Dose Level 1
Number analyzed (Participants) | 1
adverse events | 0

3. Primary Outcome: Number of Participants With a Grades 3-5 Dose-limiting Toxicity (DLT) of Continuous Intravenous (CIV) Recombinant Human Interleukin-15 (rhIL-15) Treatment
Description: A DLT is defined as a grade 3-5 toxicity if not incontrovertibly due to disease progression or an extraneous cause, and deemed possibly, probably, or definitely related to interleukin-15 by the principal investigator during the first 28 days of treatment. Some exceptions are grade 3 or 4 lymphocytopenia or neutropenia without clinical signs of infection grade 2 or above, grade 3 or 4 thrombocytopenia lasting fewer than 5 days and not associated with bleeding or purpura. Transient (<24 hours) grade 3 hypoalbuminemia, hypokalemia, hypomagnesemia, hyponatremia or hypophosphatemia which responds to medical intervention. Grade 3 is severe, grade 4 is life-threatening, and grade 5 is death related to adverse event.
Time Frame: 28 days or 4 weeks (cycle 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Dose Escalation - Dose Level 1
Number analyzed (Participants) | 1
Participants
  Grade 3 Possibly Related | 0
  Grade 3 Probably Related | 0
  Grade 3 Definitely Related | 0
  Grade 4 Possibly Related | 0
  Grade 4 Probably Related | 0
  Grade 4 Definitely Related | 0
  Grade 5 Possibly Related | 0
  Grade 5 Probably Related | 0
  Grade 5 Definitely Related | 0

4. Primary Outcome: Number of Participants With a Grade 3-5 Dose-limiting Toxicity (DLT) With Intravenous (IV) Obinutuzumab Treatment
Description: A DLT is defined as a grade 3-5 toxicity if not incontrovertibly due to disease progression or an extraneous cause, and deemed possibly, probably, or definitely related to Obinutuzumab by the principal investigator during the first 28 days of treatment. Some exceptions are grade 3 or 4 lymphocytopenia or neutropenia without clinical signs of infection grade 2 or above, grade 3 or 4 thrombocytopenia lasting fewer than 5 days and not associated with bleeding or purpura. Transient (<24 hours) grade 3 hypoalbuminemia, hypokalemia, hypomagnesemia, hyponatremia or hypophosphatemia which responds to medical intervention. Grade 3 is severe, grade 4 is life-threatening, and grade 5 is death related to adverse event.
Time Frame: 28 days or 4 weeks (cycle 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Dose Escalation - Dose Level 1
Number analyzed (Participants) | 1
Participants
  Grade 3 Possibly Related | 0
  Grade 3 Probably Related | 0
  Grade 3 Definitely Related | 0
  Grade 4 Possibly Related | 0
  Grade 4 Probably Related | 0
  Grade 4 Definitely Related | 0
  Grade 5 Possibly Related | 0
  Grade 5 Probably Related | 0
  Grade 5 Definitely Related | 0

5. Primary Outcome: Maximum Tolerated Dose (MTD) of Recombinant Human Interleukin-15 (rhIL-15) Administration
Description: The MTD is the dose level at which no more than 1 of up to 6 participants experience a dose limiting toxicity (DLT) during the DLT evaluation window, or the dose at which at least 2 of ≤ 6 participants have DLT. A DLT is defined as a grade 3-5 toxicity if not incontrovertibly due to disease progression or an extraneous cause, and deemed possibly, probably, or definitely related to interleukin-15 by the principal investigator during the first 28 days of treatment.
Time Frame: 28 days or 4 weeks (cycle 1)
Population: This outcome measure was not done. The MTD was not found because the study was closed after > 1 year of inactivity and only one participant was enrolled.
Arm/Group | Arm 1 - Dose Escalation - Dose Level 1
Number analyzed (Participants) | 0

6. Primary Outcome: Maximum Tolerated Dose (MTD) of Intravenous (IV) Obinutuzumab Treatment
Description: The MTD is the dose level at which no more than 1 of up to 6 participants experience a dose limiting toxicity (DLT) during the DLT evaluation window, or the dose at which at least 2 of ≤ 6 participants have DLT. A DLT is defined as a grade 3-5 toxicity if not incontrovertibly due to disease progression or an extraneous cause, and deemed possibly, probably, or definitely related to Obinutuzumab by the principal investigator during the first 28 days of treatment.
Time Frame: 28 days or 4 weeks (cycle 1)
Population: as for outcome 5
Arm/Group | Arm 1 - Dose Escalation - Dose Level 1
Number analyzed (Participants) | 0

7. Secondary Outcome: Duration of Response (DOR)
Description: DOR is measured from the time measurement criteria are met for complete response (CR), complete response with incomplete marrow recovery (CRi), or partial response (PR) whichever is recorded first until the first date that recurrent of progressive disease is objectively documented, death, or in the absence of progressive disease (PD), date of last assessment. Response was assessed by the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 guidelines. Complete response (CR) is disease related constitutional symptoms resolved; partial response (PR) is two criteria from Group A (e.g. lymphadenopathy or liver and/or spleen size) if abnormal at baseline plus one of the criteria from Group B (e.g. platelet count) must be met; complete response with incomplete marrow recovery (CRi) is CR with incomplete hematopoietic recovery; stable disease (SD) is defined as not achieving CR or PR, and PD is development of transformation to a more aggressive histology.
Time Frame: time measurement criteria are met for CR, CRi, or PR whichever is recorded first until the first date that recurrent of progressive disease is objectively documented or death, approximately 27 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1 - Dose Escalation - Dose Level 1
Number analyzed (Participants) | 1
Months | 0 [NA to NA] — There is no confidence interval with 1 sample result.

8. Secondary Outcome: Overall Response Rate
Description: Overall response is defined as the best response recorded from the start of the treatment until disease progression/recurrence. OS was estimated using the Kaplan-Meier curves and a 95% confidence interval. Response was assessed by the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 guidelines. Complete response (CR) is disease related constitutional symptoms resolved; Partial response (PR) is two criteria from Group A (e.g. lymphadenopathy or liver and/or spleen size) if abnormal at baseline plus one of the criteria from Group B (e.g. platelet count) must be met, requires the absence of growth factor or transfusion support; Complete response with incomplete marrow recovery (CRi) is CR with incomplete hematopoietic recovery; Stable disease (SD) is defined as not achieving CR or PR, but not fulfilling the criteria for progressive disease (PD); and PD is one criteria from Group A or B are met or development of transformation to a more aggressive histology.
Time Frame: 6 cycles (each cycle is 28 days or 4 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Dose Escalation - Dose Level 1
Number analyzed (Participants) | 1
Participants
  Complete Response | 0
  Complete Response with incomplete marrow recovery | 0
  Partial Response | 0
  Stable Disease | 1
  Progressive Disease | 0

9. Secondary Outcome: Event-free Survival (EFS)
Description: EFS is defined as the duration of time from the date of study enrollment until time of disease lapse, disease progression, alternative therapy for lymphoma given, or death, whichever comes first. EFS was estimated using the Kaplan-Meier curves and a 95% confidence interval. Progression was assessed by the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 guidelines and is defined as one criterion from Group A (e.g., lymphadenopathy or liver and/or spleen size) or B (e.g., platelet count) are met or development of transformation to a more aggressive histology.
Time Frame: Approximately 8 months
Population: There is no confidence interval with 1 sample result.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1 - Dose Escalation - Dose Level 1
Number analyzed (Participants) | 1
Months | 8

10. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the date of on-study to the date of death from any cause or last follow up.
Time Frame: Approximately 27 months
Population: There is no full range with 1 sample result.
Measure: Median (Full Range); unit: Months
Arm/Group | Arm 1 - Dose Escalation - Dose Level 1
Number analyzed (Participants) | 1
Months | 27

11. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the duration of time measurement criteria are met for complete response (CR), complete response with incomplete marrow recovery (CRi), and partial response (PR), whichever is recorded first. PFS was estimated using the Kaplan-Meier curves and a 95% confidence interval. Response was assessed by the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 guidelines. CR is disease related constitutional symptoms resolved; PR is two criteria from Group A (e.g. lymphadenopathy or liver and/or spleen size) if abnormal at baseline plus one of the criteria from Group B (e.g. platelet count) must be met, requires the absence of growth factor or transfusion support; CRi is CR with incomplete hematopoietic recovery; and progressive disease is one criteria from Group A or B are met or development of transformation to a more aggressive histology.
Time Frame: Approximately 8 months
Population: There is no full range with 1 sample result.
Measure: Median (Full Range); unit: Months
Arm/Group | Arm 1 - Dose Escalation - Dose Level 1
Number analyzed (Participants) | 1
Months | 8

12. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 27 months and 11 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Dose Escalation - Dose Level 1
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 27 months and 11 days.
Arm/Group | Arm 1 - Dose Escalation - Dose Level 1
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - Dose Escalation - Dose Level 1 (N=1)
Bone infection (Infections and infestations) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 - Dose Escalation - Dose Level 1 (N=1)
Constipation (Gastrointestinal disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2)
Paronychia (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/84/NCT03759184/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/84/NCT03759184/ICF_001.pdf